CLINICAL TRIAL: NCT02602912
Title: INJ-SPINE-01 Identification of Spine Structures by Using BIP-Needles
Brief Title: Identification of Spine Structures by Using BIP-Needles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Injeq Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: INJ-SPINE-01
Record Dates: First submitted 2015-11-09; First posted 2015-11-11 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Spinal Puncture
MeSH Terms: interventions — Needles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Injeq Bioimpedance Probe (BIP) Needle (Experimental): Injeq Bioimpedance Probe (BIP) Needle is a spinal needle that has bioimpedance measurement capability.
  Interventions: Device: Injeq Bioimpedance Probe (BIP) Needle

INTERVENTIONS:
Device: Injeq Bioimpedance Probe (BIP) Needle — Injeq Bioimpedance Probe (BIP) Needle is a spinal needle that has bioimpedance measurement capability. It consists of traditional needle cannulae and removable bioimpedance probe which enables the measurement of bioimpedance. The needle is connected to measurement device and tissue identifying algorithm. Bioimpedance is measured during the operation and the algorithm detects when the needle tip is in contact with cerebrospinal fluid.

SUMMARY:
The main purpose of the study is to assess the feasibility and clinical performance of impedance based tissue identification in various spine structures.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary adult patients going through medical operation involving spinal puncture, spinal fluid sampling or intrathecal drug injection.

Exclusion Criteria:

* Participation to other clinical study
* Exclusion criteria are the same as generally for spinal anaesthesia and lumbar punctures. Exclusion criteria includes infection on skin area, systemic anticoagulation, sepsis, anatomical unsuitability and refusal
* In addition for not giving (or not capable to give) the consent personally for any reason is an absolute exclusion criterion. In practice this means that study is for adult patients only.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
True positive and false positive detection of cerebrospinal fluid marked in case report form | During spinal puncture
  Measurement device indicates with a sound and visual feedback when needle reaches cerebrospinal fluid (CSF). Physician verifies the location by removing the needle stylet and testing whether CSF flows from the needle, similarly as in traditional process. Detection is true positive if CSF flows from the needle and false positive if not. Even if the device does not detect the spinal fluid, physician performs the CSF test when needed. Physician marks to the case report form whether the device provided detections during the spinal puncture and were the detections true or false detections.

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University Hospital, Tampere, Finland